CLINICAL TRIAL: NCT03410095
Title: The Brain Changes in Sleep Apnea Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Andrew Lim (Other)
Collaborators: University of Edinburgh (Other)
Responsible Party: Sponsor-Investigator, Dr. Andrew Lim, Scientist, staff neurologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: SleepApneaStudy
Record Dates: First submitted 2017-12-19; First posted 2018-01-25 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Sleep; Sleep Apnea; Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — Phlebotomy will be performed following an overnight fast, and samples will be banked for assessment of cytokines and endothelial biomarkers. Blood samples (45-50 ml) will be collected in plasma vacutainer tubes. Plasma will be separated and preserved in a freezer. The peripheral blood mononuclear cell (PBMC) fraction will also be kept in a freezer for genetic evaluation. All samples will be de-identified and preserved at -80oC and assayed together in a batch after the collection of the last sample (in 2020). Samples will be assayed for inflammatory and endothelial function by ELISA. Classical vascular risk factors will also be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sleep apnea patients: 80 patients recently diagnosed with severe sleep apnea will participate in the Brain Changes in Sleep Apnea Study.
  Interventions: Diagnostic Test: Brain MRI, cognitive testing, bloodwork

INTERVENTIONS:
Diagnostic Test: Brain MRI, cognitive testing, bloodwork — Participants will undergo 3-Tesla MRI. Scan time will be about 1 hour and 15 minutes per subject per session at the Sunnybrook site. The protocol is designed to image SVD burden by quantifying PVS and WMH volumes, and image various physiological estimates on the brain.
  Participants will undergo the following cognitive tests: Behavioural Neurology Assessment-R (BNA-R), Montreal Cognitive Assessment (MOCA), Center for Epidemiologic Studies Depression Scale (CES-D), and BrainScreen.
  Blood samples will be assayed for inflammatory and endothelial function. Classical vascular risk factors will also be assessed. Once data collection is complete, DNA will be extracted from the frozen PBMC fraction and will be genotyped for APOE genotype and a panel of other single nucleotide polymorphisms known to be associated with cognition and cerebrovascular disease.

SUMMARY:
Sleep is critical to human health, but insufficient and disrupted sleep caused by sleep apnea are common and have a major impact on brain health. However, there is still much that is not known about how sleep apnea damages the brain and what can be done to fix this. The Brain Changes in Sleep Apnea Study will look at the brain health of people with severe sleep apnea both before and after 4 months of treatment with a CPAP machine. Pre- and post-CPAP treatment, 80 participants with severe sleep apnea will undergo cognitive testing, blood and urine tests, a pulse wave velocity test, and an MRI. Also pre- and post-CPAP treatment, participants will wear a blood pressure monitor for 24 hours, wear an accelerometer watch for 8 nights to track the duration and quality of their sleep, and wear a device for 1 night of sleep to assess their breathing and blood oxygen levels. It is expected that there will be improvements in participants' brain health after 4 months of CPAP treatment.

DETAILED DESCRIPTION:
Between January 2018 and February 2022, the Brain Changes in Sleep Apnea Study will recruit 80 adults with newly diagnosed severe sleep apnea attending the sleep clinics at Sunnybrook Health Sciences Centre (n=40) or the University of Edinburgh (n=40). Participants will undergo home-based assessment with 3 wearable devices (24 hours of ambulatory blood pressure monitoring, 8 nights of actigraphy to assess sleep duration and fragmentation, and 1 night of finger-probe peripheral arterial tonometry and oximetry to assess cardiorespiratory physiology including sleep apnea), completion of a sleep and health questionnaire, 24-hour collection of urine for assessing sympathetic nervous system activity, blood banking for endothelial biomarkers, cognitive evaluation, pulse wave velocity test, and an MRI of the brain, at 2 time points: 1) after initial polysomnographic diagnosis of sleep apnea but before the initiation of CPAP, and 2) after 4 months of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed sleep apnea not on CPAP or any other treatment for sleep apnea;
* Apnea hypopnea index >=15 on diagnostic polysomnogram;
* Oxygen desaturation index >=10 or O2 saturation in sleep <90% for >15 minutes on diagnostic polysomnogram;
* Subjectively sleepy;
* Planning on starting CPAP for sleep apnea.

Exclusion Criteria:

* Known history of stroke, transient ischemic attack, or other CNS disease;
* Unable to safely undergo MRI;
* Use of alpha-blocking agents;
* Persistent non-sinus arrhythmia;
* Severe pulmonary or cardiac diseases including COPD and CHF;
* Waking spO2<90%;
* History of panic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 adults with newly diagnosed severe sleep apnea will be recruited from the sleep clinics at Sunnybrook Health Sciences Centre (n=40) or the University of Edinburgh (n=40).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in perivascular space volume | Baseline and 4 months
  We will use repeated measures linear mixed effect models to estimate the main effect of CPAP (i.e. compare pre- and post-CPAP measurements) on perivascular space volume.
Change from baseline in DTI fractional anisotropy on voxel-wise basis | Baseline and 4 months
  We will use repeated measures linear mixed effect models to estimate the main effect of CPAP (i.e. compare pre- and post-CPAP measurements) on DTI fractional anisotropy on voxel-wise basis.
Change from baseline in a summary measure of arterial pulsatility | Baseline and 4 months
  We will use repeated measures linear mixed effect models to estimate the main effect of CPAP (i.e. compare pre- and post-CPAP measurements) on arterial pulsatility (as measured by the pulse wave velocity test).
Change from baseline in perivascular lactate measured by MR spectroscopy | Baseline and 4 months
  We will use repeated measures linear mixed effect models to estimate the main effect of CPAP (i.e. compare pre- and post-CPAP measurements) on perivascular lactate (as measured by MR spectroscopy).
Change from baseline in cerebrovascular reactivity on a voxel-wise basis | Baseline and 4 months
  We will use repeated measures linear mixed effect models to estimate the main effect of CPAP (i.e. compare pre- and post-CPAP measurements) on cerebrovascular reactivity on a voxel-wise basis.

SECONDARY OUTCOMES:
Change from baseline in 24-hour blood pressure | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on 24-hour blood pressure (as measured by the ambulatory blood pressure monitor).
Change from baseline in sleep duration and fragmentation | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on sleep duration and fragmentation (as measured by the GENEActiv).
Change from baseline in severity of sleep apnea, % deep NREM sleep, and hypoxemia | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on severity of sleep apnea, % deep NREM sleep, and hypoxemia (as measured by the WatchPAT).
Change from baseline in serum markers of metabolic, inflammatory, cardiovascular, and endothelial function | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on serum markers of metabolic, inflammatory, cardiovascular, and endothelial function (as measured by blood tests).
Change from baseline in urinary measures of sympathetic nervous system | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on urinary measures of sympathetic nervous system (as measured with urine test).
Change from baseline in cognitive performance | Baseline and 4 months
  We will quantify the main effect of CPAP treatment on cognitive performance (as measured by our computerized battery, which includes the MoCA, BNA-R, and BrainScreen).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lim, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Ancoli-Israel S, Kripke DF, Klauber MR, Mason WJ, Fell R, Kaplan O. Sleep-disordered breathing in community-dwelling elderly. Sleep. 1991 Dec;14(6):486-95. doi: 10.1093/sleep/14.6.486. PMID 1798880
- [Background] Yaffe K, Laffan AM, Harrison SL, Redline S, Spira AP, Ensrud KE, Ancoli-Israel S, Stone KL. Sleep-disordered breathing, hypoxia, and risk of mild cognitive impairment and dementia in older women. JAMA. 2011 Aug 10;306(6):613-9. doi: 10.1001/jama.2011.1115. PMID 21828324
- [Background] Redline S, Yenokyan G, Gottlieb DJ, Shahar E, O'Connor GT, Resnick HE, Diener-West M, Sanders MH, Wolf PA, Geraghty EM, Ali T, Lebowitz M, Punjabi NM. Obstructive sleep apnea-hypopnea and incident stroke: the sleep heart health study. Am J Respir Crit Care Med. 2010 Jul 15;182(2):269-77. doi: 10.1164/rccm.200911-1746OC. Epub 2010 Mar 25. PMID 20339144
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Kim H, Yun CH, Thomas RJ, Lee SH, Seo HS, Cho ER, Lee SK, Yoon DW, Suh S, Shin C. Obstructive sleep apnea as a risk factor for cerebral white matter change in a middle-aged and older general population. Sleep. 2013 May 1;36(5):709-715B. doi: 10.5665/sleep.2632. PMID 23633753
- [Background] Lim AS, Yu L, Schneider JA, Bennett DA, Buchman AS. Sleep Fragmentation, Cerebral Arteriolosclerosis, and Brain Infarct Pathology in Community-Dwelling Older People. Stroke. 2016 Feb;47(2):516-8. doi: 10.1161/STROKEAHA.115.011608. Epub 2016 Jan 14. PMID 26768207
- [Background] Berezuk C, Ramirez J, Gao F, Scott CJ, Huroy M, Swartz RH, Murray BJ, Black SE, Boulos MI. Virchow-Robin Spaces: Correlations with Polysomnography-Derived Sleep Parameters. Sleep. 2015 Jun 1;38(6):853-8. doi: 10.5665/sleep.4726. PMID 26163465
- [Background] Malhotra A, Younes M, Kuna ST, Benca R, Kushida CA, Walsh J, Hanlon A, Staley B, Pack AI, Pien GW. Performance of an automated polysomnography scoring system versus computer-assisted manual scoring. Sleep. 2013 Apr 1;36(4):573-82. doi: 10.5665/sleep.2548. PMID 23565003
- [Background] Gottlieb DJ, Punjabi NM, Mehra R, Patel SR, Quan SF, Babineau DC, Tracy RP, Rueschman M, Blumenthal RS, Lewis EF, Bhatt DL, Redline S. CPAP versus oxygen in obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2276-85. doi: 10.1056/NEJMoa1306766. PMID 24918372
- [Background] Martinez-Garcia MA, Capote F, Campos-Rodriguez F, Lloberes P, Diaz de Atauri MJ, Somoza M, Masa JF, Gonzalez M, Sacristan L, Barbe F, Duran-Cantolla J, Aizpuru F, Manas E, Barreiro B, Mosteiro M, Cebrian JJ, de la Pena M, Garcia-Rio F, Maimo A, Zapater J, Hernandez C, Grau SanMarti N, Montserrat JM; Spanish Sleep Network. Effect of CPAP on blood pressure in patients with obstructive sleep apnea and resistant hypertension: the HIPARCO randomized clinical trial. JAMA. 2013 Dec 11;310(22):2407-15. doi: 10.1001/jama.2013.281250. PMID 24327037
- [Background] Hachinski V; World Stroke Organization. Stroke and Potentially Preventable Dementias Proclamation: Updated World Stroke Day Proclamation. Stroke. 2015 Nov;46(11):3039-40. doi: 10.1161/STROKEAHA.115.011237. No abstract available. PMID 26504189
- [Background] Kress BT, Iliff JJ, Xia M, Wang M, Wei HS, Zeppenfeld D, Xie L, Kang H, Xu Q, Liew JA, Plog BA, Ding F, Deane R, Nedergaard M. Impairment of paravascular clearance pathways in the aging brain. Ann Neurol. 2014 Dec;76(6):845-61. doi: 10.1002/ana.24271. Epub 2014 Sep 26. PMID 25204284
- [Background] Jessen NA, Munk AS, Lundgaard I, Nedergaard M. The Glymphatic System: A Beginner's Guide. Neurochem Res. 2015 Dec;40(12):2583-99. doi: 10.1007/s11064-015-1581-6. Epub 2015 May 7. PMID 25947369
- [Background] Achariyar TM, Li B, Peng W, Verghese PB, Shi Y, McConnell E, Benraiss A, Kasper T, Song W, Takano T, Holtzman DM, Nedergaard M, Deane R. Glymphatic distribution of CSF-derived apoE into brain is isoform specific and suppressed during sleep deprivation. Mol Neurodegener. 2016 Dec 8;11(1):74. doi: 10.1186/s13024-016-0138-8. PMID 27931262
- [Background] Lundblad LC, Fatouleh RH, Hammam E, McKenzie DK, Macefield VG, Henderson LA. Brainstem changes associated with increased muscle sympathetic drive in obstructive sleep apnoea. Neuroimage. 2014 Dec;103:258-266. doi: 10.1016/j.neuroimage.2014.09.031. Epub 2014 Sep 22. PMID 25255048
- [Background] Lundblad LC, Fatouleh RH, McKenzie DK, Macefield VG, Henderson LA. Brain stem activity changes associated with restored sympathetic drive following CPAP treatment in OSA subjects: a longitudinal investigation. J Neurophysiol. 2015 Aug;114(2):893-901. doi: 10.1152/jn.00092.2015. Epub 2015 May 20. PMID 25995345
- [Background] O'Brien E, Mee F, Atkins N, O'Malley K. Accuracy of the SpaceLabs 90207, Novacor DIASYS 200, Del Mar Avionics Pressurometer IV and Takeda TM-2420 ambulatory systems according to British and American criteria. J Hypertens Suppl. 1991 Dec;9(6):S332-3. No abstract available. PMID 1818987
- [Background] O'Brien E, Mee F, Atkins N, O'Malley K. Accuracy of the SpaceLabs 90207 determined by the British Hypertension Society protocol. J Hypertens. 1991 Jun;9(6):573-4. doi: 10.1097/00004872-199106000-00016. No abstract available. PMID 1653299
- [Background] Baumgart P, Kamp J. Accuracy of the SpaceLabs Medical 90217 ambulatory blood pressure monitor. Blood Press Monit. 1998 Oct;3(5):303-307. PMID 10212370
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Lichstein KL, Stone KC, Donaldson J, Nau SD, Soeffing JP, Murray D, Lester KW, Aguillard RN. Actigraphy validation with insomnia. Sleep. 2006 Feb;29(2):232-9. PMID 16494091
- [Background] Witting W, Kwa IH, Eikelenboom P, Mirmiran M, Swaab DF. Alterations in the circadian rest-activity rhythm in aging and Alzheimer's disease. Biol Psychiatry. 1990 Mar 15;27(6):563-72. doi: 10.1016/0006-3223(90)90523-5. PMID 2322616
- [Background] Sokolove PG, Bushell WN. The chi square periodogram: its utility for analysis of circadian rhythms. J Theor Biol. 1978 May 8;72(1):131-60. doi: 10.1016/0022-5193(78)90022-x. No abstract available. PMID 566361
- [Background] Sohail S, Yu L, Bennett DA, Buchman AS, Lim AS. Irregular 24-hour activity rhythms and the metabolic syndrome in older adults. Chronobiol Int. 2015;32(6):802-13. doi: 10.3109/07420528.2015.1041597. Epub 2015 Jun 10. PMID 26061588
- [Background] Lim AS, Srivastava GP, Yu L, Chibnik LB, Xu J, Buchman AS, Schneider JA, Myers AJ, Bennett DA, De Jager PL. 24-hour rhythms of DNA methylation and their relation with rhythms of RNA expression in the human dorsolateral prefrontal cortex. PLoS Genet. 2014 Nov 6;10(11):e1004792. doi: 10.1371/journal.pgen.1004792. eCollection 2014 Nov. PMID 25375876 (Retraction: PMID 34735448 PLoS Genet. 2021 Nov 4;17(11):e1009895)
- [Background] Lim AS, Yu L, Costa MD, Buchman AS, Bennett DA, Leurgans SE, Saper CB. Quantification of the fragmentation of rest-activity patterns in elderly individuals using a state transition analysis. Sleep. 2011 Nov 1;34(11):1569-81. doi: 10.5665/sleep.1400. PMID 22043128
- [Background] Lim AS, Kowgier M, Yu L, Buchman AS, Bennett DA. Sleep Fragmentation and the Risk of Incident Alzheimer's Disease and Cognitive Decline in Older Persons. Sleep. 2013 Jul 1;36(7):1027-1032. doi: 10.5665/sleep.2802. PMID 23814339
- [Background] Yalamanchali S, Farajian V, Hamilton C, Pott TR, Samuelson CG, Friedman M. Diagnosis of obstructive sleep apnea by peripheral arterial tonometry: meta-analysis. JAMA Otolaryngol Head Neck Surg. 2013 Dec;139(12):1343-50. doi: 10.1001/jamaoto.2013.5338. PMID 24158564
- [Background] Onder NS, Akpinar ME, Yigit O, Gor AP. Watch peripheral arterial tonometry in the diagnosis of obstructive sleep apnea: influence of aging. Laryngoscope. 2012 Jun;122(6):1409-14. doi: 10.1002/lary.23233. Epub 2012 Apr 20. PMID 22522750
- [Background] Hedner J, White DP, Malhotra A, Herscovici S, Pittman SD, Zou D, Grote L, Pillar G. Sleep staging based on autonomic signals: a multi-center validation study. J Clin Sleep Med. 2011 Jun 15;7(3):301-6. doi: 10.5664/JCSM.1078. PMID 21677901
- [Background] Zakzanis KK, Azarbehi R. Introducing BRAINscreen: web-based real-time examination and interpretation of cognitive function. Appl Neuropsychol Adult. 2014;21(2):77-86. doi: 10.1080/09084282.2012.742994. Epub 2013 Jun 27. PMID 24826500
- [Background] Radloff, L.S. (1977). The CED-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1, 385-401
- [Derived] Sommer R, Hill EA, Ramirez J, Coello RD, Ballerini L, Gibson E, Berberian S, Valdes Hernandez MDC, Centen A, Chappell FM, Montazeri N, Stringer MS, Thrippleton M, Jaime Garcia D, Wiseman S, Narayansingh M, Tandon A, Boulos MI, Murray BJ, Doubal F, Riha RL, Goubran M, Macintosh BJ, Wardlaw JM, Black SE, Lim ASP. Continuous Positive Airway Pressure and Progression of Enlarged Perivascular Spaces in Adults With Obstructive Sleep Apnea. Neurology. 2025 Oct;105(8):e213955. doi: 10.1212/WNL.0000000000213955. Epub 2025 Sep 29. PMID 41021868